CLINICAL TRIAL: NCT06623929
Title: Evaluation of Topical Analgesia Treatments for Ankle Sprains
Brief Title: Topical Treatments for Ankle Sprains
Status: Active, not recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Elif Kaya Çelikel, MD, Ankara City Hospital Bilkent
Other Study IDs: AEŞH-EK1-2023-750
Record Dates: First submitted 2024-09-12; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Ankle Sprain
Keywords: local anesthesia; emergency; Nonsteroidal Anti-Inflammatory Drug; Ankle sprain
MeSH Terms: conditions — Ankle Injuries; Emergencies | interventions — Diclofenac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group E: Group E, Etofenamate spray 100 mg/ml (Flexo 100 mg/ml-Kocaeli) is applied to the painful area from a distance of approximately 10-15 cm in a maximum of 7 puffs. Each puff contains 18 mg etofenamate.
  Interventions: Drug: Etofenamat
- Group D: Group D Diclofenac diethylammonium 1% spray (Painout Ice 1%-Ankara) was applied to the painful area from a distance of approximately 10-15 cm in a maximum of 6 puffs. Each puff contained 5.8 mg diclofenac diethylammonium.
  Interventions: Drug: Diclofenac

INTERVENTIONS:
Drug: Etofenamat — E group: Etofenamate spray 100 mg/ml is applied to the painful area from a distance of approximately 10-15 cm in a maximum of 7 puffs. Each puff contains 18 mg etofenamate.
  Groups: Group E
Drug: Diclofenac — Group D: Diclofenac diethylammonium 1% spray was applied to the painful area from a distance of approximately 10-15 cm in a maximum of 6 puffs. Each puff contained 5.8 mg diclofenac diethylammonium.
  Groups: Group D

SUMMARY:
Our aim was to evaluate the effects of topical analgesic drugs on rapid recovery of joint functions and pain relief in acute ankle injuries.

A total of 100 patients were included in the study and divided into 2 groups as Diclofenac and Etofenamate. The pain scores of the patients were evaluated with the Numeric Rating scale and Wong-Baker scale before and after treatment. Dorsiflexion and plantarflexion active joint movements were measured with a hand-held goniometer for joint function before and after treatment.

We found that ankle sprains were more common in men. In our study, we found that both topical analgesics were effective in improving joint movements and reducing pain.

ELIGIBILITY:
Inclusion Criteria:Those over the age of 18, who applied to the emergency room within the first 48 hours after an ankle sprain, who have grade 1/mild and grade 2/moderate ankle sprains, who have excluded fractures and dislocations, who have no muscle-tendon ruptures, no vascular or nerve injuries, no open wounds or burns, whose vital signs are stable, and who give written and verbal consent.

-

Exclusion Criteria:Those who did not present within the first 48 hours of ankle sprain, grade 3/severe ankle sprain, multiple trauma, pregnancy, suspected pregnancy, foot and ankle fractures and dislocations, those who had a previous ankle operation or fracture, and cases who did not accept to participate in the study

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases presenting to the emergency department with an ankle sprain within the first 48 hours
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Drugs and Pain | 0., 1. hour
  It is the recovery of pain, swelling in the acute phase of ankle sprain.

SECONDARY OUTCOMES:
Drugs and movement | 0., and 1. hour
  It is the recovery of joint movement functions in the acute phase of ankle sprain.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Ankara, Turkey (Türkiye)